CLINICAL TRIAL: NCT01388764
Title: Pilot Study: To Assess the Safety, Tolerability and Effects of L-Arginine on Muscles in Boys With Dystrophinopathy on Corticosteroids
Brief Title: Safety, Tolerability and Effects of L-Arginine in Boys With Dystrophinopathy on Corticosteroids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Namita Goyal, Physician Neurologist, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2011D001591
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Dystrophinopathy; Duchenne Muscular Dystrophy; Becker's Muscular Dystrophy
Keywords: L-arginine supplement study
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-arginine (Experimental)
  Interventions: Drug: L-arginine

INTERVENTIONS:
Drug: L-arginine — Subjects will receive oral L-Arginine (0.3 grams/kg/day, divided 2 times per day, not to exceed 14 grams/day)

SUMMARY:
The purpose of the study is to assess the safety, tolerability, and effects of L-Arginine on muscles in boys with dystrophinopathy on corticosteroids. Specifically, to see if L-arginine reduces muscle signal abnormalities on MRI done pre and post 30 days of L-arginine administration.

DETAILED DESCRIPTION:
Dystrophinopathy is a muscular dystrophy (includes Duchenne or Becker's Muscular Dystrophy) that can be a lethal muscle disorder resulting from defects in the gene for dystrophin, a structural protein required to maintain muscle integrity. Absence of functional dystrophin leaves the muscle membrane vulnerable to damage during contraction. This damage can be exacerbated by an inflammatory response leading to myofiber necrosis.

L-arginine is a widely available dietary supplement amino acid postulated to affect dystrophinopathy in several favorable ways: upregulation of utrophin, vasodilation in muscle via nitric oxide, enhanced synthesis of creatine, increase levels of growth hormone.

We hypothesize that administration of L-arginine may increase levels of creatine and growth hormone and in turn reduce the extent of myofiber damage in our patients with dystrophinopathy

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of diagnosis of dystrophinopathy, documented by clinical exam and dystrophin DNA mutation analysis
* Ambulatory male subjects between the ages of 7-11 years
* Stable dosage of corticosteroids for 3 months prior to entry (Screening/Baseline Day 0) and during treatment period
* Able to follow instructions and give assent
* Able to complete nonsedated MR

Exclusion Criteria:

* Presence of metallic orthopedic hardware in the lower extremity that could affect MRI/MRS measurements
* Routine MRI exclusion criteria such as the presence of a pacemaker, cochlear implant, or cerebral aneurysm clip
* Subjects not capable of cooperating during MR examination
* Known hypersensitivity to L-arginine
* Exposure to another investigational agent, investigational supplements, growth hormone within 3 months prior to entry (Screening/Baseline Day 0) or during treatment period
* Subjects must not be taking L-arginine for at least 4 weeks prior to entry (Day 0)
* Subjects who are non-ambulatory or with daytime ventilatory dependence

Ages: 7 Years to 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
MRI/MRS of calf muscle | Day 0 and Day 30
  MRI/MRS will be performed of the calf muscle in all subjects (N=8) to assess muscle signal abnormalities on MRI and creatine levels on MRS, done at the start of the study (Day 0) and at the end of the study (Day 30), after 30 days of L-arginine administration.

SECONDARY OUTCOMES:
Blood tests | Day 0 and Day 30
  We will obtain safety labs [complete blood count (CBC) and comprehensive metabolic panel (CMP)] from all subjects (N =8), at day 0 and day 30, after 30 days of oral L-argninine administration.
Assessment of muscle strength and function | Day 0 and Day 30
  Measurements of upper and lower extremity strength will be performed using a hand-held dynamometer. Functional tests will also be performed which include time to walk specified distances and time to climb stairs.
Pulmonary function tests | Day 0 and Day 30
  Subjects will have pulmonary function studies to assess forced vital capacity

CONTACTS AND LOCATIONS:
Overall Officials: Namita Goyal, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States